CLINICAL TRIAL: NCT03563313
Title: A Pivotal Study of t:Slim X2 With Control-IQ Technology
Brief Title: The International Diabetes Closed Loop (iDCL) Trial: Clinical Acceptance of the Artificial Pancreas
Acronym: DCLP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Jaeb Center for Health Research (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry); Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DCLP3; UC4DK108483 (NIH)
Record Dates: First submitted 2018-06-07; First posted 2018-06-20 (Actual); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas (AP); Type 1 Diabetes Mellitus; Insulin Pump; Continuous Glucose Monitor (CGM); Closed Loop Control (CLC); Sensor-Augmented Pump (SAP)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of 6 month at home closed loop system vs. sensor-augmented pump.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Closed Loop Control (CLC) (Experimental): Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 6 months.
  Interventions: Device: t:slim X2 with Control-IQ Technology & Dexcom G6 CGM
- Sensor-Augmented Pump (SAP) (Active Comparator): Participants randomized to sensor-augmented pump (SAP) will use an insulin pump with no automated insulin delivery and a study CGM (Dexcom G6) for 6 months.
  Interventions: Device: Sensor-augmented pump (SAP)

INTERVENTIONS:
Device: t:slim X2 with Control-IQ Technology & Dexcom G6 CGM — Participants will use the Tandem t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 6 months at home.
  Arms: Closed Loop Control (CLC)
Device: Sensor-augmented pump (SAP) — Participants will use an insulin pump with no automated insulin delivery and a study CGM (Dexcom G6) for 6 months at home. Pump-users at the time of enrollment will use their personal pump in this arm. Multiple daily injection (MDI) users at the time of enrollment will use a t:slim X2 insulin pump without Control-IQ technology.
  Arms: Sensor-Augmented Pump (SAP)

SUMMARY:
The objective of the study is to assess efficacy and safety of a closed loop system (t:slim X2 with Control-IQ Technology) in a large randomized controlled trial.

DETAILED DESCRIPTION:
After consent is signed, eligibility will be assessed. Eligible participants not currently using an insulin pump and Dexcom CGM with minimum data requirements will initiate a run-in phase of 2 to 8 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 2:1 to the use of closed-loop control (CLC group) using t:slim X2 with Control-IQ Technology vs. SAP for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year.
2. Familiarity and use of a carbohydrate ratio for meal boluses.
3. Age ≥14.0 years old.
4. For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
5. For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact the participant in case of an emergency.
6. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use.
7. Willingness to use a regular insulin pump during the study with no automatic insulin adjustment based on glucose level when assigned to participate in an SAP group
8. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
9. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study.
10. Total daily insulin dose (TDD) at least 10 U/day.
11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.

Exclusion Criteria

1. Concurrent use of any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
2. Hemophilia or any other bleeding disorder.
3. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk.
4. Participation in another pharmaceutical or device trial at the time of enrollment or during the study.
5. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc. or TypeZero Technologies, LLC, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue A. Brown, MD, Principal Investigator — University of Virginia
Locations (7):
- United States (7):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - Harvard University (Joslin Diabetes Center), Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally, data will be made available after the primary publications of each study.
Access Criteria: The Data Sharing Agreements will be formulated by the Steering Committee in collaboration with the NIH Project Scientist Program Official.
  In addition, under special arrangements, complete data sets will be provided to industry partners who would use the data for regulatory clearance (PMA - pre-market approval) of the tested artificial pancreas system. This will be done in response to the specific requirements of RFA-DK-14-024 for this project to "…generate data able to satisfy safety and efficacy requirements by regulatory agencies regarding the clinical testing of artificial pancreas device systems" in the target population of people with type 1 diabetes.

REFERENCES:
- [Derived] Beck RW, Kanapka LG, Breton MD, Brown SA, Wadwa RP, Buckingham BA, Kollman C, Kovatchev B. A Meta-Analysis of Randomized Trial Outcomes for the t:slim X2 Insulin Pump with Control-IQ Technology in Youth and Adults from Age 2 to 72. Diabetes Technol Ther. 2023 May;25(5):329-342. doi: 10.1089/dia.2022.0558. Epub 2023 Apr 12. PMID 37067353
- [Derived] Kanapka LG, Lum JW, Beck RW. Insulin Pump Infusion Set Failures Associated with Prolonged Hyperglycemia: Frequency and Relationship to Age and Type of Infusion Set During 22,741 Infusion Set Wears. Diabetes Technol Ther. 2022 Jun;24(6):396-402. doi: 10.1089/dia.2021.0548. Epub 2022 Feb 23. PMID 35104166
- [Derived] Ekhlaspour L, Town M, Raghinaru D, Lum JW, Brown SA, Buckingham BA. Glycemic Outcomes in Baseline Hemoglobin A1C Subgroups in the International Diabetes Closed-Loop Trial. Diabetes Technol Ther. 2022 Aug;24(8):588-591. doi: 10.1089/dia.2021.0524. Epub 2022 Feb 8. PMID 35020488
- [Derived] Kudva YC, Laffel LM, Brown SA, Raghinaru D, Pinsker JE, Ekhlaspour L, Levy CJ, Messer LH, Kovatchev BP, Lum JW, Beck RW, Gonder-Frederick L; iDCL Trial Research Group. Patient-Reported Outcomes in a Randomized Trial of Closed-Loop Control: The Pivotal International Diabetes Closed-Loop Trial. Diabetes Technol Ther. 2021 Oct;23(10):673-683. doi: 10.1089/dia.2021.0089. PMID 34115959
- [Derived] Isganaitis E, Raghinaru D, Ambler-Osborn L, Pinsker JE, Buckingham BA, Wadwa RP, Ekhlaspour L, Kudva YC, Levy CJ, Forlenza GP, Beck RW, Kollman C, Lum JW, Brown SA, Laffel LM; iDCL Trial Research Group. Closed-Loop Insulin Therapy Improves Glycemic Control in Adolescents and Young Adults: Outcomes from the International Diabetes Closed-Loop Trial. Diabetes Technol Ther. 2021 May;23(5):342-349. doi: 10.1089/dia.2020.0572. Epub 2021 Jan 21. PMID 33216667
- [Derived] O'Malley G, Messer LH, Levy CJ, Pinsker JE, Forlenza GP, Isganaitis E, Kudva YC, Ekhlaspour L, Raghinaru D, Lum J, Brown SA; iDCL Trial Research Group. Clinical Management and Pump Parameter Adjustment of the Control-IQ Closed-Loop Control System: Results from a 6-Month, Multicenter, Randomized Clinical Trial. Diabetes Technol Ther. 2021 Apr;23(4):245-252. doi: 10.1089/dia.2020.0472. PMID 33155824
- [Derived] Brown SA, Kovatchev BP, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, Laffel LM, Levy CJ, Pinsker JE, Wadwa RP, Dassau E, Doyle FJ 3rd, Anderson SM, Church MM, Dadlani V, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Kollman C, Beck RW; iDCL Trial Research Group. Six-Month Randomized, Multicenter Trial of Closed-Loop Control in Type 1 Diabetes. N Engl J Med. 2019 Oct 31;381(18):1707-1717. doi: 10.1056/NEJMoa1907863. Epub 2019 Oct 16. PMID 31618560

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Started | 112 | 56
Completed | 112 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP) | Total
Number analyzed (Participants) | 112 | 56 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 17 | 48
  Between 18 and 65 years | 81 | 39 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (16) | 33 (17) | 33 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 30 | 84
  Male | 58 | 26 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 18
  Not Hispanic or Latino | 99 | 51 | 150
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 0 | 4
  White | 94 | 53 | 147
  More than one race | 7 | 1 | 8
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 112 | 56 | 168
CGM Time in Target Range 70-180 mg/dL [Mean (Standard Deviation); unit: percentage of time] — CGM percentage of time in target range measured over 2-week baseline.
  percentage of time | 61 (17) | 59 (14) | 60 (16)

OUTCOME MEASURES:

1. Primary Outcome: Time in Target Range
Description: The primary outcome is time in target range 70-180 mg/dL measured by CGM in CLC group vs. SAP group.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage of time | 71 (12) | 59 (14)
Statistical Analysis 1: Comparison: Closed Loop Control (CLC) vs Sensor-Augmented Pump (SAP); Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: CGM Time Above 180
Description: CGM-measured % above 180 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 27 (12) | 38 (15)
Statistical Analysis 1: Comparison: Closed Loop Control (CLC) vs Sensor-Augmented Pump (SAP); Test type: Superiority; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: CGM Mean Glucose
Description: CGM-measured mean glucose
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
mg/dL | 156 (19) | 170 (25)
Statistical Analysis 1: Comparison: Closed Loop Control (CLC) vs Sensor-Augmented Pump (SAP); Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: HbA1c at 26 Weeks
Description: Hemoglobin A1c measured at 26 weeks
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 7.06 (0.79) | 7.39 (0.92)
Statistical Analysis 1: Comparison: Closed Loop Control (CLC) vs Sensor-Augmented Pump (SAP); Test type: Superiority; p = 0.001, Mixed Models Analysis

5. Secondary Outcome: CGM Time Below 70
Description: CGM-measured % below 70 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 1.58 (1.15) | 2.25 (1.46)
Statistical Analysis 1: Comparison: Closed Loop Control (CLC) vs Sensor-Augmented Pump (SAP); Test type: Superiority; p < 0.001, Mixed Models Analysis

6. Secondary Outcome: CGM Time Below 54
Description: CGM-measured % below 54 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 0.29 (0.29) | 0.35 (0.32)
Statistical Analysis 1: Comparison: Closed Loop Control (CLC) vs Sensor-Augmented Pump (SAP); Test type: Superiority; p = 0.02, Mixed Models Analysis

7. Secondary Outcome: CGM Time in Range 70-140 mg/dL
Description: CGM-measured % in range 70-140 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 46 (12) | 36 (12)

8. Secondary Outcome: Coefficient of Variability
Description: CGM measured glucose variability measured with the coefficient of variation (CV)
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage SD of Mean
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage SD of Mean | 34 (5) | 36 (5)

9. Secondary Outcome: Standard Deviation of CGM
Description: CGM measured glucose variability measured with the standard deviation (SD)
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
mg/dL | 53 (12) | 62 (13)

10. Secondary Outcome: CGM Time Below 60
Description: CGM-measured % below 60 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 0.58 (0.52) | 0.75 (0.61)

11. Secondary Outcome: LBGI
Description: Low blood glucose index by CGM with higher index indicating higher risk of hypoglycemia. Values <1 suggest minimal risk. Index of risk of low blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale (Kovatchev BP, Cox DJ, Gonder-Frederick LA, Young-Hyman D, Schlundt D, Clarke WL: Assessment of risk for severe hypoglycemia among adults with IDDM: validation of the low blood glucose index. Diabetes Care 21:1870-1875, 1998)
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
units on a scale | 0.51 (0.29) | 0.65 (0.35)

12. Secondary Outcome: CGM Hypoglycemia Events
Description: CGM-measured events of at least 15 consecutive minutes <70mg/dL per week
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
events per week | 3.3 (2.1) | 4.3 (2.7)

13. Secondary Outcome: CGM Time >250
Description: CGM-measured % >250 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 7 (6.7) | 12.3 (10.2)

14. Secondary Outcome: CGM Time >300
Description: CGM-measured % >300 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 2.4 (3.4) | 4.6 (6.0)

15. Secondary Outcome: HBGI
Description: High blood glucose index by CGM with higher values indicating higher risk of hyperglycemia. Index of risk of high blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale (Kovatchev BP, Cox DJ, Kumar A, Gonder-Frederick L, Clarke WL. Algorithmic evaluation of metabolic control and risk of severe hypoglycemia in type 1 and type 2 diabetes using self-monitoring blood glucose data. Diabetes Technol Ther 2003;5:817-828pmid:14633347)
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
index | 6.3 (3.1) | 9.0 (4.4)

16. Secondary Outcome: Number of Participants With HbA1c <7.0% at 26 Weeks
Description: Number of participants HbA1c <7.0% at 26 weeks
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
Participants | 52 | 17

17. Secondary Outcome: Number of Participants With HbA1c <7.5% at 26 Weeks
Description: Number of Participants with HbA1c <7.5% at 26 weeks
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
Participants | 79 | 33

18. Secondary Outcome: Number of Participants With HbA1c Improvement From Baseline to 26 Weeks >0.5%
Description: HbA1c improvement from baseline to 26 weeks >0.5%
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 35 | 6

19. Secondary Outcome: Number of Participants With HbA1c Improvement From Baseline to 26 Weeks >1.0%
Description: HbA1c improvement from baseline to 26 weeks >1.0%
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 12 | 0

20. Secondary Outcome: HbA1c Relative Improvement From Baseline to 26 Weeks >10%
Description: HbA1c relative improvement from baseline to 26 weeks >10%
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
percentage | 21 (19) | 2 (4)

21. Secondary Outcome: Number of Participants With HbA1c Improvement From Baseline to 26 Weeks >1.0% or HbA1c <7.0% at 26 Weeks
Description: HbA1c improvement from baseline to 26 weeks >1.0% or HbA1c <7.0% at 26 weeks
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 59 | 17

22. Secondary Outcome: HFS-II
Description: For adults, teens and parents items on this survey are rated on a 5 point Likert scale from never (0) to almost always (4). The survey is scored by summing item responses. Fear of Hypoglycemia Survey (HFS-II) for adults has a total score that is summed from the two subscale scores (33 items) and ranges from 0 to 132 with higher scores indicating greater degrees of fear of hypoglycemia. The teen survey has a total of 25 items and the range of Total scores is 0 to 100. The parent version of the survey has a total of 26 items with Total scores that range from 0 to 108.
Time Frame: 26 weeks
Population: Total Score at 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Closed Loop Control (CLC) in Adults: Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 6 months.
  t:slim X2 with Control-IQ Technology & Dexcom G6 CGM: Participants will use the Tandem t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 6 months at home.
- Sensor-Augmented Pump (SAP) in Adults: Participants randomized to sensor-augmented pump (SAP) will use an insulin pump with no automated insulin delivery and a study CGM (Dexcom G6) for 6 months.
  Sensor-augmented pump (SAP): Participants will use an insulin pump with no automated insulin delivery and a study CGM (Dexcom G6) for 6 months at home. Pump-users at the time of enrollment will use their personal pump in this arm. Multiple daily injection (MDI) users at the time of enrollment will use a t:slim X2 insulin pump without Control-IQ technology.
- CLC in Teens: Survey response from a teen in CLC (14-18 years old)
- SAP in Teens: Survey response from a Teen in the SAP group (ages 14-18).
- Parent of Teen in CLC: Survey response from a parent of a teen in CLC
- Parent of a Teen in SAP: Survey response from a parent of a teen in SAP
Arm/Group | Closed Loop Control (CLC) in Adults | Sensor-Augmented Pump (SAP) in Adults | CLC in Teens | SAP in Teens | Parent of Teen in CLC | Parent of a Teen in SAP
Number analyzed (Participants) | 80 | 39 | 31 | 16 | 31 | 15
score on a scale | 33 (12) | 38 (18) | 32 (10) | 31 (16) | 33 (14) | 36 (15)

23. Secondary Outcome: Hyperglycemia Avoidance Scale
Description: Hyperglycemia Avoidance Scale total score is the sum of 21 items rated on a 4 point Likert scale from 0 (never) to 4 (almost always) and ranges from 0 to 84 with a higher score indicating greater degrees of avoiding hyperglycemia.
Time Frame: 26 weeks
Population: Total Score at 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
score on a scale | 39 (7) | 37 (11)

24. Secondary Outcome: Diabetes Distress Scale
Description: Diabetes Distress Scale for adults has 28 items rated on a 6 point Likert scale that ranges from 1 (not a problem) to 6 (a very serious problem). The total score is the mean of the sum of responses and ranges from 1 to 6 where a higher score indicates greater degrees of diabetes distress.
Time Frame: 26 weeks
Population: Total Score at 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
score on a scale | 1.7 (0.6) | 1.9 (0.8)

25. Secondary Outcome: Hypoglycemia Confidence Scale
Description: Hypoglycemia Confidence Scale has 20 items which are rated on a 4-point Likert Scale ranging from 1 (not confident at all) to 4 (very confident) with higher scores indicating higher confidence in dealing with hypoglycemia. A single score is computed by calculating the mean of the sum of all items and ranges from 1 to 4.
Time Frame: 26 weeks
Population: First two items on hypoglycemia confidence scale
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Closed Loop Control (CLC) in Adults | Sensor-Augmented Pump (SAP) in Adults
Number analyzed (Participants) | 111 | 55
score on a scale
  Execise | 2.3 [0 to 3] | 1.9 [0 to 3]
  Sleeping | 2.3 [1 to 3] | 1.9 [0 to 3]

26. Secondary Outcome: Clarke Hypoglycemia Awareness Scores
Description: Clarke Hypoglycemia Awareness Scores (0-7 score with higher scores associated with impaired awareness)
Time Frame: 26 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
score on a scale | 1 [0 to 3] | 2 [0 to 3]

27. Secondary Outcome: INSPIRE Survey Scores
Description: The INSPIRE questionnaire assesses user expectations and experiences with Insulin Delivery Systems: Perceptions, Ideas, Reflections, Expectations (INSPIRE). Survey total scores are computed by calculating the mean of the sum of all item ratings then multiplying the mean by 25 to scale the score to a range from 0 to 100. Higher scores indicate a more positive perception of insulin delivery systems. Items are rated on a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The Adult survey has 22 items, the Teens/Adolescents survey has 17 items and the Parent survey has 21 items.
Time Frame: 26 weeks
Population: Scores are measured at 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed Loop Control (CLC) in Adults | Sensor-Augmented Pump (SAP) in Adults | CLC in Teens | SAP in Teens | Parent of Teen in CLC | Parent of a Teen in SAP
Number analyzed (Participants) | 80 | 39 | 31 | 16 | 31 | 15
score on a scale | 87 (14) | 86 (13) | 87 (13) | 74 (12) | 87 (13) | 76 (12)

28. Secondary Outcome: System Usability Scores (SUS)
Description: System Usability Scores (SUS)-composite score from 0 to 100 with higher scores indicate better perceived usability
Time Frame: 26 weeks
Population: Administered to CLC group only. Results from 26-week.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed Loop Control (CLC)
Number analyzed (Participants) | 109
score on a scale | 87 (12)

29. Secondary Outcome: Technology Acceptance Questionnaire
Description: Technology Acceptance Survey measures the user's perceptions regarding the burdens and the barriers associated with a technology with a higher score indicates increased technology acceptance. There total score uses 37 items with items are rated on a 5 point scale ranging from 1 (strongly disagree) to 5 (strongly agree) for total score range of 37-185.
Time Frame: 26 weeks
Population: Administered to CLC arm only. Result from 26-weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed Loop Control (CLC)
Number analyzed (Participants) | 111
score on a scale | 155 (19)

30. Secondary Outcome: Total Daily Insulin
Description: Total Daily Insulin (units)
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
units | 55 (27) | 51 (20)

31. Secondary Outcome: Basal:Bolus Insulin Ratio
Description: Basal:Bolus Insulin Ratio
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
ratio | 1.1 (0.7) | 1.1 (0.8)

32. Secondary Outcome: Weight
Description: Weight (kg)
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
kilograms | 78.7 (17.0) | 76.0 (18.9)

33. Secondary Outcome: BMI
Description: Body Mass Index (BMI) kg/m^2
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 111 | 55
kg/m^2 | 26.2 (4.9) | 26.1 (6.1)

34. Other Pre Specified Outcome: Number of Participants With Severe Hypoglycemia (Per Protocol)
Description: Severe hypoglycemia (per protocol)
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 0 | 0

35. Other Pre Specified Outcome: Number of Participants With Diabetic Ketoacidosis (Per Protocol)
Description: Diabetic ketoacidosis (per protocol)
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 1 | 0

36. Other Pre Specified Outcome: Ketone Events Defined as Day With Ketone Level >1.0 mmol/L
Description: Ketone events defined as day with ketone level >1.0 mmol/L
Time Frame: 26 weeks
Measure: Number; unit: days
Units Other Than Participants: Days
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Number analyzed (Days) | 20571 | 10285
days | 14 | 15

37. Other Pre Specified Outcome: CGM-measured Hypoglycemic Events (>15 Minutes With Glucose Concentration <54 mg/dL)
Description: CGM-measured hypoglycemic events (>15 minutes with glucose concentration <54 mg/dL)
Time Frame: 26 weeks
Measure: Median (Inter-Quartile Range); unit: events per week
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
events per week | 0.4 [0.1 to 0.9] | 0.5 [0.2 to 0.9]

38. Other Pre Specified Outcome: CGM-measured Hyperglycemic Events (>15 Minutes With Glucose Concentration >300 mg/dL)
Description: CGM-measured hyperglycemic events (>15 minutes with glucose concentration >300 mg/dL)
Time Frame: 26 weeks
Measure: Median (Inter-Quartile Range); unit: events per week
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
events per week | 1.2 [0.4 to 2.6] | 2.7 [1.1 to 4.6]

39. Other Pre Specified Outcome: BG-measured Hypoglycemic Events (One BG Record <54 mg/dL)
Description: BG-measured hypoglycemic events (one BG record <54 mg/dL)
Time Frame: 26 weeks
Measure: Number; unit: days
Units Other Than Participants: Days
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Number analyzed (Days) | 20571 | 10285
days | 129 | 72

40. Other Pre Specified Outcome: BG-measured Hyperglycemic Events (One BG Record >350 mg/dL)
Description: BG-measured hyperglycemic events (one BG record >350 mg/dL)
Time Frame: 26 weeks
Measure: Number; unit: days
Units Other Than Participants: Days
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Number analyzed (Days) | 20571 | 10285
days | 243 | 181

41. Other Pre Specified Outcome: Worsening of HbA1c From Baseline to 26 Weeks by >0.5%
Description: Worsening of HbA1c from baseline to 26 weeks by >0.5%
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 8 | 5

42. Other Pre Specified Outcome: Other Serious Adverse Events (SAE) and Serious Adverse Device Events (SADE)
Description: Other serious adverse events (SAE) and serious adverse device events (SADE)
Time Frame: 26 weeks
Population: Other Serious Adverse Events that do not include DKA or Severe Hypoglycemia
Measure: Number; unit: participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
participants
  Concussion | 1 | 0
  Otitis | 1 | 0
  Cardiac Bypass Surgery | 1 | 0

43. Other Pre Specified Outcome: Adverse Device Effects (ADE)
Description: Adverse device effects (ADE)
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) in Adults | Sensor-Augmented Pump (SAP) in Adults
Number analyzed (Participants) | 112 | 56
Participants | 11 | 0

44. Other Pre Specified Outcome: Unanticipated Adverse Device Effects (UADE)
Description: Unanticipated adverse device effects (UADE)
Time Frame: 26 weeks
Population: Study Device
Measure: Number; unit: Unanticipated Adverse Device Effects
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Unanticipated Adverse Device Effects | 1 | 0

45. Other Pre Specified Outcome: Number of Participants With SH Events
Description: For this outcome, mean +/- SD or summary statistics appropriate to the distribution will be tabulated by treatment group
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 0 | 0

46. Other Pre Specified Outcome: SH Event Rate Per 100 Person-years
Description: For this outcome, severe hypoglycemia event rate per 100 person-years will be calculated as a rate.
Time Frame: 26 weeks
Measure: Number; unit: rate per 100 person-years
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
rate per 100 person-years | 0 | 0

47. Other Pre Specified Outcome: Number of Participants With DKA Events
Description: For this outcome, number of participants with diabetic ketoacidosis (DKA) will be tabulated.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
Participants | 1 | 0

48. Other Pre Specified Outcome: DKA Event Rate Per 100 Person-years
Description: For this outcome, the diabetic ketoacidosis event rate per 100 person-years will be calculated as a rate.
Time Frame: 26 weeks
Measure: Number; unit: rate per 100 person-years
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
rate per 100 person-years | 1.8 | 0

49. Other Pre Specified Outcome: Any Adverse Event Rate Per 100 Person-years
Description: For this outcome, the adverse event rate per 100 person-years calculated as a rate.
Time Frame: 26 weeks
Measure: Number; unit: events per 100 person-yr
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 112 | 56
events per 100 person-yr | 30.2 | 7.1

ADVERSE EVENTS:
Time Frame: From protocol entry through last study date which is approximately 26-28 weeks per participant.
Description: Definitions are the same as the clinicaltrials.gov definition. Please see clinical protocol for exclusions to adverse event collection.
Arm/Group | Closed Loop Control (CLC) | Sensor-Augmented Pump (SAP)
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/56
Serious Adverse Events (participants affected / at risk) | 4/112 | 0/56
Other Adverse Events (participants affected / at risk) | 12/112 | 2/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Loop Control (CLC) (N=112) | Sensor-Augmented Pump (SAP) (N=56)
Diabetic Ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 1 (1) | 0 (0)
Otitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cardiac Bypass Surgery (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Loop Control (CLC) (N=112) | Sensor-Augmented Pump (SAP) (N=56)
Hyperglycemia or ketosis events without meeting criteria for Diabetic Ketoacidosis (Endocrine disorders) | 12 (13) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT03563313/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03563313/SAP_001.pdf
  • Informed Consent Form (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT03563313/ICF_002.pdf